CLINICAL TRIAL: NCT05226169
Title: Randomized Controlled Trial of Intravenous Ferric Carboxymaltose for Iron-Deficiency Anemia in Patients With Advanced Gastric Cancer Receiving Palliative Chemotherapy
Brief Title: Efficacy and Safety oF FErric CarboxymalTose in Patients With Advanced Gastric Cancer(EFFECT-AGC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC2102
Record Dates: First submitted 2021-12-27; First posted 2022-02-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Advanced Gastric Carcinoma
MeSH Terms: interventions — ferric carboxymaltose; Fosfomycin; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment arm : IV FCM (Experimental): Intravenous ferric carboxymaltose
  Interventions: Drug: Ferinject
- Control treatment arm: Conservative management (Active Comparator): Conservative management
  * Absolute IDA: oral ferrous sulfate
  * Functional IDA: no treatment or oral ferrous sulfate according to the physician's choice
  * Other IV iron or PRC transfusion or ESA therapy is not allowed
  Interventions: Other: Conservative management

INTERVENTIONS:
Drug: Ferinject — * Patients will receive an IV FCM (1,000 mg iron) infusion on the first day (visit 1) of chemotherapy. FCM (FerinjectTM; Vifor Pharma, Glattbrugg, Switzerland) will be diluted in 250 ml of sterile 0.9% normal saline by an aseptic technique and infused over 15 min under the supervision of a clinician.
  * Patients with a Hb level ≤ 10 g/dL and ID (serum ferritin < 100 ng/mL or TSAT < 50% and serum ferritin 100-500 ng/mL) will receive an additional dose of 500 mg of IV FCM at 6, 12, 24, 36, and 48 weeks. FCM will be diluted in 100 ml of sterile 0.9% normal saline by an aseptic technique and infused over 6 min under the supervision of a clinician.
  Other Names: IV FCM
  Arms: Active treatment arm : IV FCM
Other: Conservative management — * Patients with absolute (must be administered) or functional (according to the physician's choice) IDA in the control arm will be received oral iron, administered as Feroba-You 256mg once or twice a day. Advice will be given regarding ingestion without food and with liquid high in ascorbic acid to maximize enteric absorption.
  * If patients in the control arm still meet the absolute or functional IDA at the end of study (at 48 weeks), they can receive IV FCM (1,000 mg) according to the physician's decision.
  Arms: Control treatment arm: Conservative management

SUMMARY:
The main objective of this study is to evaluate the efficacy and safety of IV FCM(ferric carboxymaltose) in patients with AGC receiving palliative chemotherapy. This study will also evaluate the effect of IV FCM on the treatment outcomes of palliative chemotherapy in patients with gastric cancer receiving fluoropyrimidine and platinum-based regimen in the same 1st-line palliative setting.

DETAILED DESCRIPTION:
Gastric cancer is associated with chronic blood loss, poor nutrition, and surgical interventions interfering with iron absorption, all of which synergistically increase the risk of iron-deficiency anemia (IDA). A retrospective review of gastric cancer reported that at the time of gastric cancer diagnosis, the prevalence of anemia was 58.7% and the overall prevalence of IDA was 40%. Moreover, patients with unresectable locally advanced or metastatic gastric cancer are treated with myelosuppressive chemotherapies, which further increases the risk for anemia.

The absorption of oral iron in gastric cancer patients is limited due to malabsorption, ongoing gastrointestinal bleeding, and lack of adherence to treatment due to dyspepsia, vomiting, abdominal pain, diarrhea, and constipation. Therefore, IV iron may be preferable due to easy administration, effective iron absorption, and infrequent complications in gastric cancer patients.

• There are a number of IV iron formulations in the market; the recommended IV iron preparations are low-molecular-weight iron dextran, ferric gluconate, iron sucrose, ferric carboxymaltose (FCM), and ferumoxytol. FCM (FerinjectTM; Vifor Pharma, Glattbrugg, Switzerland) is a stable colloidal solution of nanoparticles which consist of a polynuclear iron (III)-(oxyhydr)oxide core stabilized by carboxymaltose, which allows slow and prolonged iron release, and is given as a single high-dose (1,000 mg of iron) in a 15-minute infusion. Based on extensive experience in clinical trial and real-world settings, IV FCM is an effective and generally well tolerated treatment for rapidly replenishing iron stores and correcting anemia in patients with ID or IDA of various etiologies.

FCM was effective in patients with active malignancy and IDA (n=420), and hematological malignancies or solid tumors and anemia (n=367) in two real-world, noninterventional studies conducted in Germany and France. Recently, two prospective studies conducted in South Korea have reported a significant increase in Hb levels by treatment with IV FCM in patients with solid cancers (including gastric cancer) receiving chemotherapy and in patients with acute isovolemic anemia following gastrectomy.

Therefore, the main objective of this study is to evaluate the efficacy and safety of IV FCM in patients with AGC receiving palliative chemotherapy. This study will also evaluate the effect of IV FCM on the treatment outcomes of palliative chemotherapy in patients with gastric cancer receiving fluoropyrimidine and platinum-based regimen in the same 1st-line palliative setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years at the time of study registration
2. Eastern Cooperative Oncology Group performance status ≤ 2
3. Histologically or cytologically confirmed gastric or gastroesophageal junction (GEJ) adenocarcinoma
4. Locally advanced unresectable or metastatic disease
5. Patients who have not been treated with palliative systemic antitumor agents for advanced or recurrent gastric or GEJ adenocarcinoma
6. Patients scheduled to receive palliative first-line fluoropyrimidine and platinum-based systemic therapy including targeted therapy or immunotherapy
7. Life expectancy ≥24 weeks
8. IDA

   1. Hb 8 to <11 g/dL
   2. Absolute ID (serum ferritin < 100 ng/mL) OR functional ID (TSAT* < 50% and serum ferritin 100-500 ng/mL)

      * TSAT = (serum iron level x 100)/ total iron-binding capacity (TIBC)

Exclusion Criteria:

1. Body weight < 35 kg
2. Immediate need for transfusion or Hb < 8 g/dL
3. Possible functional ID or No ID (serum ferritin > 500 ng/mL OR TSAT ≥ 50%)
4. Anemia attributable to factors other than cancer or chemotherapy (e.g., vitamin B12 and/or serum folate deficiency; hemolysis; or myelodysplastic syndromes)
5. Ongoing bleeding or overt gross active bleeding (e.g., hematemesis, melena, or hematochezia)
6. Neoplastic bone marrow infiltration
7. History of ESA, IV or oral iron therapy, and/or RBC transfusion 4 weeks prior to randomization
8. Iron overload or disturbances in utilization of iron (e.g., personal or family history of hemochromatosis and hemosiderosis)
9. Known hypersensitivity to any of the required study products or known serious hypersensitivity to other parenteral iron products
10. Known severe allergies including drug allergies, history of severe asthma, eczema or other atopic allergies, and in subjects with immune or inflammatory conditions (e.g., systemic lupus erythematosus, rheumatoid arthritis)
11. Decreased renal function including renal dialysis (previous, current or planned within the next 6 months,) or serum creatinine levels ≥ 2.0 mg/dL, or estimated glomerular filtration rate < 30 mL/min/1.73 m2
12. Chronic liver disease (including active hepatitis) and/or aspartate transaminase (AST) or alanine transaminase (ALT) ≥ 3 times the upper limit of the normal range
13. Active acute or chronic infections (assessed by clinical judgment)
14. Other significant medical condition(s) in the opinion of the investigator with an anticipated need for major surgery during the study, or any other kind of disorder that may be associated with increased risk to the subject or may interfere with study assessments, outcomes (e.g., uncontrolled hypertension, active cardiac disease, thromboembolic disease, or uncontrolled diabetes mellitus, neurological or psychiatric disorders)
15. Pregnancy (e.g., positive human chorionic gonadotropin test) or breast-feeding. If the subject is of childbearing potential and does, not use adequate contraceptive precautions. The subject must agree to use adequate contraception during the study and for 1 month after the last dose of study treatment. A highly effective method of birth control must be used.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum change of Hb concentration | baseline to 12 weeks
  Maximum change of Hb concentration from baseline to 12 weeks (or first RBC transfusion and/or ESA, or study withdrawl, or death, whichever will be first) without RBC transfusion and/or ESA

SECONDARY OUTCOMES:
Change of Hb concentration | baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
  Change of Hb concentration from baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
Change in serum iron | baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
  Change in serum iron from baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
Change in serum ferritin | baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
  Change in serum iron, ferritin(ng/dL) from baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
Change in serum TIBC | baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
  Change in serum TIBC(µg/dL) from baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
Change in serum TSAT | baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
  Change in serum TSAT(%) from baseline to 3, 6, 9, 12, 24, 36, and 48 weeks
Tumor response | every 6-8weeks, assessed up to 24 months
  according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  time from the date of first administration of palliative first-line chemotherapy to the date of the first objectively documented tumor progression or death, whichever occurs first)
OS | through study completion, an average of 2 years
  time from the date of first administration of palliative first-line chemotherapy to the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided